CLINICAL TRIAL: NCT00999466
Title: A Double-blind, Placebo-controlled, Randomised, Parallel Group, Phase IIa Study to Investigate the Efficacy, Tolerability and Safety of 8 Doses of AZD8848 Administered Intranasally Once Weekly in Mild to Moderate Allergic Asthma Subjects Challenged With an Inhaled Allergen.
Brief Title: The Tolerability and Effects of AZD8848 in Allergic Asthma Subjects Challenged With Inhaled Allergen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0540C00004
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Results first posted 2016-01-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Allergic Asthma
MeSH Terms: interventions — AZD8848

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD8848 (30 μg PILOT part and 60 μg MAIN part)
  Interventions: Drug: AZD8848
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8848 — Nasal spray, solution 0.6mg/ mL. Once weekly for 7 weeks, 8 doses in total.
  Arms: 1
Drug: Placebo — Nasal spray, solution. Once weekly for 7 weeks, 8 doses in total.
  Arms: 2

SUMMARY:
AZD8848 is a new drug that is being tested for the treatment of asthma and allergic rhinitis (hayfever). This study will be in two parts and will include 59 asthmatic patients in total. The first part will investigate the tolerability and safety of AZD8848 while the second part will investigate both the therapeutic effect of AZD8848 and how well patients tolerate the drug.

ELIGIBILITY:
Inclusion Criteria:

* FEV1 > 70 % of predicted normal pre-bronchodilator
* Documented history of asthma
* Presence of allergic sensitivity

Exclusion Criteria:

* Clinically relevant disease and/or abnormality (past or present), which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results of the study, or the patient's ability to participate in the study.
* Symptomatic allergic rhinitis
* Any clinical relevant abnormal findings in physical examination or assessment which may put the patient at risk because of participation in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10; Primary Completion 2011-02 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leif Eriksson, MD, Study Director — AstraZeneca R&D Lund; Brian Leaker, MD, Principal Investigator — Respiratory Clinical Trials
Locations (2):
- United Kingdom (2):
  - Research Site, London
  - Research Site, Manchester

REFERENCES:
- [Derived] Leaker BR, Singh D, Lindgren S, Almqvist G, Eriksson L, Young B, O'Connor B. Effects of the Toll-like receptor 7 (TLR7) agonist, AZD8848, on allergen-induced responses in patients with mild asthma: a double-blind, randomised, parallel-group study. Respir Res. 2019 Dec 19;20(1):288. doi: 10.1186/s12931-019-1252-2. PMID 31856838
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=191&filename=D0540C00004_Study_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD8848, 30 μg: AZD8848 nasal spray, 30 μg, one spray in the left nostril once weekly. Pilot part.
- AZD8848, 60 μg: AZD8848 nasal spray, 60 μg, one spray of 30 μg per nostril once weekly. Main part.
- Placebo: Placebo nasal spray, one spray in the left nostril (Pilot part) or per nostril (Main part) once weekly.
Period: Pilot Part
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Started | 6 | 0 (AZD8848 nasal spray 60 μg group was not participated in the Pilot part) | 3
Completed | 6 | 0 | 3
Not Completed | 0 | 0 | 0
Period: Main Part
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Started | 0 (AZD8848 nasal spray 30 μg group was not participated in the Main part) | 26 | 25
Completed | 0 | 22 | 21
Not Completed | 0 | 4 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Adverse Event | 0 | 4 | 2

BASELINE CHARACTERISTICS:
Population: AZD8848 30 μg nasal spray was only done in Pilot part. 3 of the 28 placebo subjects were from the PILOT part and 25 placebo subjects were from the MAIN part.
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo | Total
Number analyzed (Participants) | 6 | 26 | 28 | 60
Age, Continuous [Mean (Full Range); unit: Years] | 36.3 [23 to 47] | 33.0 [19 to 51] | 32.3 [21 to 50] | 33.9 [19 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 7 | 7 | 14
  Male | 6 | 19 | 21 | 46

OUTCOME MEASURES:

1. Primary Outcome: FEV1, Late Asthmatic Response (LAR) - Pre-treatment
Description: Forced Expiratory Volume in 1 second (FEV1), Late Asthmatic Response (LAR), is derived as the ratio of FEV1 Area Under Curve 4-10 hour post allergen challenge (AUC 4-10h) (computed using the trapezoidal formula divided by time) and the pre-challenge FEV1 measurement.
Time Frame: Pre-treatment (Baseline measurement)
Population: There were 6 AZD8848 nasal spray 30 μg subjects and 3 placebo subjects participated in the Pilot part only that they did not have outcome measure collected. The number of participants analyzed for each outcome measure were subset of the subjects who participated in the Main part and also provided data for that measure.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 22 | 23
ratio |  | 0.814 (0.450) | 1.01 (0.784)

2. Primary Outcome: FEV1, Late Asthmatic Response (LAR) - 1 Week After Last Dose
Description: FEV1, Late Asthmatic Response (LAR), is derived as the ratio of FEV1 AUC 4-10h (computed using the trapezoidal formula divided by time) and the pre-challenge FEV1 measurement.
Time Frame: 1 week after last dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 22 | 23
ratio |  | 0.616 (0.296) | 0.970 (0.641)

3. Primary Outcome: FEV1, Late Asthmatic Response (LAR) - 4 Weeks After Last Dose
Description: as for outcome 2
Time Frame: 4 weeks after last dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 22 | 21
ratio |  | 0.759 (0.397) | 0.722 (0.584)

4. Secondary Outcome: FEV1, Early Asthmatic Response (EAR) - Pre-treatment
Description: FEV1, Early Asthmatic Response (EAR), is derived as the ratio of FEV1 Area Under Curve 0-2 hour post allergen challenge (AUC 0-2h) (computed using the trapezoidal formula divided by time) and the pre-challenge FEV1 measurement.
Time Frame: Pre-treatment (Baseline measurement)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 22 | 23
ratio |  | 0.524 (0.241) | 0.611 (0.362)

5. Secondary Outcome: FEV1, Early Asthmatic Response (EAR) - 1 Week After Last Dose
Description: FEV1, Early Asthmatic Response (EAR), is derived as the ratio of FEV1 AUC 0-2h (computed using the trapezoidal formula divided by time) and the pre-challenge FEV1 measurement.
Time Frame: 1 week after last dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 22 | 23
ratio |  | 0.468 (0.361) | 0.624 (0.362)

6. Secondary Outcome: FEV1, Early Asthmatic Response (EAR) - 4 Weeks After Last Dose
Description: as for outcome 5
Time Frame: 4 weeks after last dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 22 | 21
ratio |  | 0.510 (0.240) | 0.591 (0.401)

7. Secondary Outcome: PC20 Methacholine Challenge - Pre-treatment, Pre Allergen Challenge
Description: PC20 is the provocation concentration of Methacholine causing a 20% fall in FEV1
Time Frame: Pre-treatment, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: mg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 22 | 23
mg/mL |  | 0.564 [0.004 to 11.1] | 0.609 [0.063 to 5.69]

8. Secondary Outcome: PC20 Methacholine Challenge - Pre-treatment, Post Allergen Challenge
Description: PC20 is the provocation concentration of Methacholine causing a 20% fall in FEV1
Time Frame: Pre-treatment, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: mg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 22 | 23
mg/mL |  | 0.425 [0.123 to 6.25] | 0.364 [0.063 to 10.2]

9. Secondary Outcome: PC20 Methacholine Challenge - 1 Week After Last Dose, Pre Allergen Challenge
Description: PC20 is the provocation concentration of Methacholine causing a 20% fall in FEV1
Time Frame: 1 week after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: mg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 22 | 21
mg/mL |  | 0.488 [0.063 to 3.01] | 0.454 [0.063 to 8.25]

10. Secondary Outcome: PC20 Methacholine Challenge - 1 Week After Last Dose, Post Allergen Challenge
Description: PC20 is the provocation concentration of Methacholine causing a 20% fall in FEV1
Time Frame: 1 week after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: mg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 21 | 21
mg/mL |  | 0.691 [0.063 to 9.13] | 0.340 [0.063 to 17.8]

11. Secondary Outcome: PC20 Methacholine Challenge - 4 Weeks After Last Dose, Pre Allergen Challenge
Description: PC20 is the provocation concentration of Methacholine causing a 20% fall in FEV1
Time Frame: 4 weeks after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: mg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 22 | 21
mg/mL |  | 0.468 [0.063 to 2.47] | 0.504 [0.072 to 4.00]

12. Secondary Outcome: PC20 Methacholine Challenge - 4 Weeks After Last Dose, Post Allergen Challenge
Description: PC20 is the provocation concentration of Methacholine causing a 20% fall in FEV1
Time Frame: 4 weeks after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: mg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 21 | 20
mg/mL |  | 0.326 [0.082 to 4.08] | 0.508 [0.063 to 29.1]

13. Secondary Outcome: Sputum Cellularity and Cytokines, Tumour Necrosis Factor Alpha (TNFα) - Pre-treatment, Pre Allergen Challenge
Time Frame: Pre-treatment, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 12 | 19
pg/mL |  | 8.9 [3.5 to 25] | 4.8 [0.90 to 24]

14. Secondary Outcome: Sputum Cellularity and Cytokines, TNFα - Pre-treatment, Post Allergen Challenge
Time Frame: Pre-treatment, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
pg/mL |  | 13 [2.8 to 156] | 12 [5.3 to 38]

15. Secondary Outcome: Sputum Cellularity and Cytokines, TNFα - 1 Week After Last Dose, Pre Allergen Challenge
Time Frame: 1 week after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 19
pg/mL |  | 6.5 [1.7 to 46] | 5.3 [0.90 to 23]

16. Secondary Outcome: Sputum Cellularity and Cytokines, TNFα - 1 Week After Last Dose, Post Allergen Challenge
Time Frame: 1 week after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
pg/mL |  | 11 [2.4 to 539] | 8.4 [1.1 to 41]

17. Secondary Outcome: Sputum Cellularity and Cytokines, TNFα - 4 Weeks After Last Dose, Pre Allergen Challenge
Time Frame: 4 weeks after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 17
pg/mL |  | 5.1 [0.90 to 113] | 9.4 [1.5 to 510]

18. Secondary Outcome: Sputum Cellularity and Cytokines, TNFα - 4 Weeks After Last Dose, Post Allergen Challenge
Time Frame: 4 weeks after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 13 | 16
pg/mL |  | 13 [4.3 to 125] | 7.9 [4.4 to 23]

19. Secondary Outcome: Sputum Cellularity and Cytokines, Interleukin-1β (IL-1β) - Pre-treatment, Pre Allergen Challenge
Time Frame: Pre-treatment, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 12 | 19
pg/mL |  | 37 [6.5 to 127] | 23 [0.80 to 243]

20. Secondary Outcome: Sputum Cellularity and Cytokines, IL-1β - Pre-treatment, Post Allergen Challenge
Time Frame: Pre-treatment, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
pg/mL |  | 41 [13 to 322] | 44 [13 to 320]

21. Secondary Outcome: Sputum Cellularity and Cytokines, IL-1β - 1 Week After Last Dose, Pre Allergen Challenge
Time Frame: 1 week after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 19
pg/mL |  | 37 [7.8 to 614] | 36 [4.5 to 139]

22. Secondary Outcome: Sputum Cellularity and Cytokines, IL-1β - 1 Week After Last Dose, Post Allergen Challenge
Time Frame: 1 week after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
pg/mL |  | 45 [7.0 to 293] | 37 [13 to 217]

23. Secondary Outcome: Sputum Cellularity and Cytokines, IL-1β - 4 Weeks After Last Dose, Pre Allergen Challenge
Time Frame: 4 weeks after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 17
pg/mL |  | 29 [6.6 to 303] | 43 [7.6 to 366]

24. Secondary Outcome: Sputum Cellularity and Cytokines, IL-1β - 4 Weeks After Last Dose, Post Allergen Challenge
Time Frame: 4 weeks after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 13 | 16
pg/mL |  | 72 [15 to 198] | 41 [15 to 224]

25. Secondary Outcome: Sputum Cellularity and Cytokines, Interleukin-5 (IL-5) - Pre-treatment, Pre Allergen Challenge
Time Frame: Pre-treatment, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 12 | 19
pg/mL |  | 0.83 [0.40 to 9.0] | 0.87 [0.40 to 5.6]

26. Secondary Outcome: Sputum Cellularity and Cytokines, IL-5 - Pre-treatment, Post Allergen Challenge
Time Frame: Pre-treatment, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
pg/mL |  | 7.1 [0.40 to 74] | 5.8 [0.40 to 27]

27. Secondary Outcome: Sputum Cellularity and Cytokines, IL-5 - 1 Week After Last Dose, Pre Allergen Challenge
Time Frame: 1 week after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 19
pg/mL |  | 0.82 [0.40 to 4.5] | 1.3 [0.40 to 11]

28. Secondary Outcome: Sputum Cellularity and Cytokines, IL-5 - 1 Week After Last Dose, Post Allergen Challenge
Time Frame: 1 week after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
pg/mL |  | 7.8 [1.1 to 38] | 5.4 [0.90 to 35]

29. Secondary Outcome: Sputum Cellularity and Cytokines, IL-5 - 4 Weeks After Last Dose, Pre Allergen Challenge
Time Frame: 4 weeks after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 17
pg/mL |  | 1.2 [0.40 to 5.5] | 1.7 [0.40 to 24]

30. Secondary Outcome: Sputum Cellularity and Cytokines, IL-5 - 4 Weeks After Last Dose, Post Allergen Challenge
Time Frame: 4 weeks after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 13 | 16
pg/mL |  | 5.7 [0.80 to 38] | 8.0 [2.1 to 47]

31. Secondary Outcome: Sputum Cellularity and Cytokines, Interleukin-6 (IL-6) - Pre-treatment, Pre Allergen Challenge
Time Frame: Pre-treatment, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 12 | 19
pg/mL |  | 15 [4.4 to 61] | 9.4 [0.40 to 189]

32. Secondary Outcome: Sputum Cellularity and Cytokines, IL-6 - Pre-treatment, Post Allergen Challenge
Time Frame: Pre-treatment, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
pg/mL |  | 28 [5.7 to 252] | 27 [1.7 to 75]

33. Secondary Outcome: Sputum Cellularity and Cytokines, IL-6 - 1 Week After Last Dose, Pre Allergen Challenge
Time Frame: 1 week after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 19
pg/mL |  | 15 [2.4 to 43] | 9.6 [0.40 to 37]

34. Secondary Outcome: Sputum Cellularity and Cytokines, IL-6 - 1 Week After Last Dose, Post Allergen Challenge
Time Frame: 1 week after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
pg/mL |  | 26 [5.2 to 142] | 23 [3.1 to 76]

35. Secondary Outcome: Sputum Cellularity and Cytokines, IL-6 - 4 Weeks After Last Dose, Pre Allergen Challenge
Time Frame: 4 weeks after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 17
pg/mL |  | 12 [0.60 to 123] | 21 [6.3 to 1317]

36. Secondary Outcome: Sputum Cellularity and Cytokines, IL-6 - 4 Weeks After Last Dose, Post Allergen Challenge
Time Frame: 4 weeks after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 13 | 16
pg/mL |  | 20 [5.3 to 174] | 29 [10 to 107]

37. Secondary Outcome: Sputum Cellularity and Cytokines, Interleukin-8 (IL-8) - Pre-treatment, Pre Allergen Challenge
Time Frame: Pre-treatment, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 12 | 19
pg/mL |  | 766 [138 to 1784] | 522 [8.5 to 2500]

38. Secondary Outcome: Sputum Cellularity and Cytokines, IL-8 - Pre-treatment, Post Allergen Challenge
Time Frame: Pre-treatment, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
pg/mL |  | 1300 [422 to 2500] | 1450 [549 to 2500]

39. Secondary Outcome: Sputum Cellularity and Cytokines, IL-8 - 1 Week After Last Dose, Pre Allergen Challenge
Time Frame: 1 week after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 19
pg/mL |  | 720 [186 to 2500] | 609 [63 to 2366]

40. Secondary Outcome: Sputum Cellularity and Cytokines, IL-8 - 1 Week After Last Dose, Post Allergen Challenge
Time Frame: 1 week after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
pg/mL |  | 1272 [284 to 2500] | 1270 [240 to 2500]

41. Secondary Outcome: Sputum Cellularity and Cytokines, IL-8 - 4 Weeks After Last Dose, Pre Allergen Challenge
Time Frame: 4 weeks after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 17
pg/mL |  | 496 [68 to 2500] | 1012 [176 to 2500]

42. Secondary Outcome: Sputum Cellularity and Cytokines, IL-8 - 4 Weeks After Last Dose, Post Allergen Challenge
Time Frame: 4 weeks after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 13 | 16
pg/mL |  | 1500 [783 to 2500] | 1304 [595 to 2500]

43. Secondary Outcome: Sputum Cellularity and Cytokines, Interleukin-10 (IL-10) - Pre-treatment, Pre Allergen Challenge
Time Frame: Pre-treatment, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 12 | 19
pg/mL |  | 0.57 [0.50 to 1.1] | 0.63 [0.50 to 2.6]

44. Secondary Outcome: Sputum Cellularity and Cytokines, IL-10 - Pre-treatment, Post Allergen Challenge
Time Frame: Pre-treatment, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
pg/mL |  | 0.86 [0.50 to 32] | 0.68 [0.50 to 1.7]

45. Secondary Outcome: Sputum Cellularity and Cytokines, IL-10 - 1 Week After Last Dose, Pre Allergen Challenge
Time Frame: 1 week after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 19
pg/mL |  | 0.60 [0.50 to 2.5] | 0.75 [0.50 to 34]

46. Secondary Outcome: Sputum Cellularity and Cytokines, IL-10 - 1 Week After Last Dose, Post Allergen Challenge
Time Frame: 1 week after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
pg/mL |  | 0.79 [0.50 to 53] | 0.82 [0.50 to 3.0]

47. Secondary Outcome: Sputum Cellularity and Cytokines, IL-10 - 4 Weeks After Last Dose, Pre Allergen Challenge
Time Frame: 4 weeks after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 17
pg/mL |  | 0.54 [0.50 to 0.90] | 0.95 [0.50 to 17]

48. Secondary Outcome: Sputum Cellularity and Cytokines, IL-10 - 4 Weeks After Last Dose, Post Allergen Challenge
Time Frame: 4 weeks after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 13 | 16
pg/mL |  | 0.68 [0.50 to 1.9] | 0.67 [0.50 to 5.7]

49. Secondary Outcome: Sputum Cellularity and Cytokines, Interleukin-13 (IL-13) - Pre-treatment, Pre Allergen Challenge
Time Frame: Pre-treatment, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 12 | 19
pg/mL |  | 1.3 [1.2 to 3.6] | 1.4 [1.2 to 3.8]

50. Secondary Outcome: Sputum Cellularity and Cytokines, IL-13 - Pre-treatment, Post Allergen Challenge
Time Frame: Pre-treatment, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
pg/mL |  | 3.0 [1.2 to 25] | 3.1 [1.2 to 9.2]

51. Secondary Outcome: Sputum Cellularity and Cytokines, IL-13 - 1 Week After Last Dose, Pre Allergen Challenge
Time Frame: 1 week after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 19
pg/mL |  | 1.3 [1.2 to 1.9] | 1.8 [1.2 to 8.0]

52. Secondary Outcome: Sputum Cellularity and Cytokines, IL-13 - 1 Week After Last Dose, Post Allergen Challenge
Time Frame: 1 week after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
pg/mL |  | 3.0 [1.2 to 8.3] | 2.8 [1.2 to 20]

53. Secondary Outcome: Sputum Cellularity and Cytokines, IL-13 - 4 Weeks After Last Dose, Pre Allergen Challenge
Time Frame: 4 weeks after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 17
pg/mL |  | 1.3 [1.2 to 2.1] | 1.6 [1.2 to 6.5]

54. Secondary Outcome: Sputum Cellularity and Cytokines, IL-13 - 4 Weeks After Last Dose, Post Allergen Challenge
Time Frame: 4 weeks after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 13 | 16
pg/mL |  | 2.5 [1.2 to 11] | 3.1 [1.2 to 17]

55. Secondary Outcome: Sputum Cellularity and Cytokines, Total Cells/g - Pre-treatment, Pre Allergen Challenge
Time Frame: Pre-treatment, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: Cell count/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 12 | 19
Cell count/g |  | 2.7 [1.3 to 6.8] | 2.7 [0.67 to 14]

56. Secondary Outcome: Sputum Cellularity and Cytokines, Total Cells/g - Pre-treatment, Post Allergen Challenge
Time Frame: Pre-treatment, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: Cell count/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
Cell count/g |  | 5.0 [1.1 to 35] | 3.5 [0.25 to 7.9]

57. Secondary Outcome: Sputum Cellularity and Cytokines, Total Cells/g - 1 Week After Last Dose, Pre Allergen Challenge
Time Frame: 1 week after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: Cell count/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 19
Cell count/g |  | 3.7 [0.84 to 16] | 3.0 [0.95 to 20]

58. Secondary Outcome: Sputum Cellularity and Cytokines, Total Cells/g - 1 Week After Last Dose, Post Allergen Challenge
Time Frame: 1 week after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: Cell count/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
Cell count/g |  | 5.0 [1.9 to 19] | 4.2 [0.55 to 18]

59. Secondary Outcome: Sputum Cellularity and Cytokines, Total Cells/g - 4 Weeks After Last Dose, Pre Allergen Challenge
Time Frame: 4 weeks after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: Cell count/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 16
Cell count/g |  | 1.9 [0.29 to 9.4] | 2.6 [0.58 to 12]

60. Secondary Outcome: Sputum Cellularity and Cytokines, Total Cells/g - 4 Weeks After Last Dose, Post Allergen Challenge
Time Frame: 4 weeks after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: Cell count/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 13 | 16
Cell count/g |  | 5.2 [2.2 to 15] | 4.0 [1.2 to 12]

61. Secondary Outcome: Sputum Cellularity and Cytokines, Eosinophils - Pre-treatment, Pre Allergen Challenge
Time Frame: Pre-treatment, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 12 | 19
10^6 cells/g |  | 0.13 [0.015 to 0.46] | 0.12 [0.008 to 3.7]

62. Secondary Outcome: Sputum Cellularity and Cytokines, Eosinophils - Pre-treatment, Post Allergen Challenge
Time Frame: Pre-treatment, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
10^6 cells/g |  | 0.64 [0.008 to 6.5] | 0.81 [0.023 to 3.0]

63. Secondary Outcome: Sputum Cellularity and Cytokines, Eosinophils - 1 Week After Last Dose, Pre Allergen Challenge
Time Frame: 1 week after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 19
10^6 cells/g |  | 0.18 [0.033 to 2.1] | 0.23 [0.008 to 2.8]

64. Secondary Outcome: Sputum Cellularity and Cytokines, Eosinophils - 1 Week After Last Dose, Post Allergen Challenge
Time Frame: 1 week after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
10^6 cells/g |  | 0.94 [0.12 to 3.8] | 0.82 [0.066 to 6.0]

65. Secondary Outcome: Sputum Cellularity and Cytokines, Eosinophils - 4 Weeks After Last Dose, Pre Allergen Challenge
Time Frame: 4 weeks after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 16
10^6 cells/g |  | 0.13 [0.009 to 2.2] | 0.21 [0.032 to 1.1]

66. Secondary Outcome: Sputum Cellularity and Cytokines, Eosinophils - 4 Weeks After Last Dose, Post Allergen Challenge
Time Frame: 4 weeks after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 13 | 16
10^6 cells/g |  | 1.0 [0.20 to 5.8] | 0.96 [0.13 to 4.6]

67. Secondary Outcome: Sputum Cellularity and Cytokines, Neutrophils - Pre-treatment, Pre Allergen Challenge
Time Frame: Pre-treatment, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 12 | 19
10^6 cells/g |  | 0.75 [0.026 to 4.2] | 0.93 [0.026 to 10]

68. Secondary Outcome: Sputum Cellularity and Cytokines, Neutrophils - Pre-treatment, Post Allergen Challenge
Time Frame: Pre-treatment, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
10^6 cells/g |  | 1.9 [0.45 to 25] | 1.5 [0.061 to 4.1]

69. Secondary Outcome: Sputum Cellularity and Cytokines, Neutrophils - 1 Week After Last Dose, Pre Allergen Challenge
Time Frame: 1 week after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 19
10^6 cells/g |  | 1.5 [0.065 to 15] | 0.91 [0.026 to 17]

70. Secondary Outcome: Sputum Cellularity and Cytokines, Neutrophils - 1 Week After Last Dose, Post Allergen Challenge
Time Frame: 1 week after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
10^6 cells/g |  | 2.1 [0.36 to 9.1] | 1.7 [0.22 to 15]

71. Secondary Outcome: Sputum Cellularity and Cytokines, Neutrophils - 4 Weeks After Last Dose, Pre Allergen Challenge
Time Frame: 4 weeks after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 16
10^6 cells/g |  | 0.80 [0.097 to 7.5] | 1.3 [0.072 to 9.3]

72. Secondary Outcome: Sputum Cellularity and Cytokines, Neutrophils - 4 Weeks After Last Dose, Post Allergen Challenge
Time Frame: 4 weeks after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 13 | 16
10^6 cells/g |  | 2.6 [0.81 to 11] | 1.6 [0.40 to 7.8]

73. Secondary Outcome: Sputum Cellularity and Cytokines, Macrophages - Pre-treatment, Pre Allergen Challenge
Time Frame: Pre-treatment, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 12 | 19
10^6 cells/g |  | 1.1 [0.29 to 2.2] | 0.59 [0.004 to 3.7]

74. Secondary Outcome: Sputum Cellularity and Cytokines, Macrophages - Pre-treatment, Post Allergen Challenge
Time Frame: Pre-treatment, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
10^6 cells/g |  | 1.1 [0.13 to 4.9] | 0.60 [0.10 to 2.1]

75. Secondary Outcome: Sputum Cellularity and Cytokines, Macrophages - 1 Week After Last Dose, Pre Allergen Challenge
Time Frame: 1 week after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 19
10^6 cells/g |  | 0.80 [0.088 to 3.1] | 0.36 [0.004 to 2.4]

76. Secondary Outcome: Sputum Cellularity and Cytokines, Macrophages - 1 Week After Last Dose, Post Allergen Challenge
Time Frame: 1 week after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
10^6 cells/g |  | 1.0 [0.20 to 5.2] | 0.77 [0.12 to 3.0]

77. Secondary Outcome: Sputum Cellularity and Cytokines, Macrophages - 4 Weeks After Last Dose, Pre Allergen Challenge
Time Frame: 4 weeks after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 16
10^6 cells/g |  | 0.47 [0.004 to 1.9] | 0.58 [0.22 to 1.6]

78. Secondary Outcome: Sputum Cellularity and Cytokines, Macrophages - 4 Weeks After Last Dose, Post Allergen Challenge
Time Frame: 4 weeks after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 13 | 16
10^6 cells/g |  | 0.56 [0.087 to 1.8] | 0.74 [0.083 to 4.0]

79. Secondary Outcome: Sputum Cellularity and Cytokines, Lymphocytes - Pre-treatment, Pre Allergen Challenge
Time Frame: Pre-treatment, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 12 | 19
10^6 cells/g |  | 0.004 [0.002 to 0.027] | 0.004 [0.002 to 0.059]

80. Secondary Outcome: Sputum Cellularity and Cytokines, Lymphocytes - Pre-treatment, Post Allergen Challenge
Time Frame: Pre-treatment, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
10^6 cells/g |  | 0.008 [0.002 to 0.086] | 0.004 [0.002 to 0.060]

81. Secondary Outcome: Sputum Cellularity and Cytokines, Lymphocytes - 1 Week After Last Dose, Pre Allergen Challenge
Time Frame: 1 week after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 19
10^6 cells/g |  | 0.002 [0.002 to 0.016] | 0.003 [0.002 to 0.046]

82. Secondary Outcome: Sputum Cellularity and Cytokines, Lymphocytes - 1 Week After Last Dose, Post Allergen Challenge
Time Frame: 1 week after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
10^6 cells/g |  | 0.003 [0.002 to 0.040] | 0.003 [0.002 to 0.045]

83. Secondary Outcome: Sputum Cellularity and Cytokines, Lymphocytes - 4 Weeks After Last Dose, Pre Allergen Challenge
Time Frame: 4 weeks after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 16
10^6 cells/g |  | 0.005 [0.002 to 0.035] | 0.005 [0.002 to 0.036]

84. Secondary Outcome: Sputum Cellularity and Cytokines, Lymphocytes - 4 Weeks After Last Dose, Post Allergen Challenge
Time Frame: 4 weeks after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 13 | 16
10^6 cells/g |  | 0.005 [0.002 to 0.049] | 0.003 [0.002 to 0.012]

85. Secondary Outcome: Sputum Cellularity and Cytokines, Epithelial Cells - Pre-treatment, Pre Allergen Challenge
Time Frame: Pre-treatment, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 12 | 19
10^6 cells/g |  | 0.045 [0.001 to 0.29] | 0.053 [0.001 to 0.59]

86. Secondary Outcome: Sputum Cellularity and Cytokines, Epithelial Cells - Pre-treatment, Post Allergen Challenge
Time Frame: Pre-treatment, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
10^6 cells/g |  | 0.078 [0.001 to 3.5] | 0.073 [0.001 to 0.35]

87. Secondary Outcome: Sputum Cellularity and Cytokines, Epithelial Cells - 1 Week After Last Dose, Pre Allergen Challenge
Time Frame: 1 week after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 19
10^6 cells/g |  | 0.11 [0.008 to 0.39] | 0.045 [0.001 to 1.4]

88. Secondary Outcome: Sputum Cellularity and Cytokines, Epithelial Cells - 1 Week After Last Dose, Post Allergen Challenge
Time Frame: 1 week after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 17 | 17
10^6 cells/g |  | 0.067 [0.001 to 0.56] | 0.071 [0.001 to 0.47]

89. Secondary Outcome: Sputum Cellularity and Cytokines, Epithelial Cells - 4 Weeks After Last Dose, Pre Allergen Challenge
Time Frame: 4 weeks after last dose, pre allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 16 | 16
10^6 cells/g |  | 0.045 [0.005 to 0.20] | 0.054 [0.001 to 0.43]

90. Secondary Outcome: Sputum Cellularity and Cytokines, Epithelial Cells - 4 Weeks After Last Dose, Post Allergen Challenge
Time Frame: 4 weeks after last dose, post allergen challenge
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 10^6 cells/g
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Number analyzed (Participants) | 0 | 13 | 16
10^6 cells/g |  | 0.037 [0.001 to 0.17] | 0.082 [0.018 to 0.24]

ADVERSE EVENTS:
Arm/Group | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 0 | 0 | 1
Other Adverse Events (participants affected / at risk) | 6 | 22 | 24
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
Tonsillitis Bacterial (Infections and infestations) | 0/6 | 0/26 | 1/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | AZD8848, 30 μg | AZD8848, 60 μg | Placebo
TINNITUS (Ear and labyrinth disorders) | 1/6 | 0/26 | 1/28
Eye Pruritus (Eye disorders) | 0/6 | 0/26 | 2/28
LACRIMATION INCREASED (Eye disorders) | 0/6 | 0/26 | 2/28
EYE SWELLING (Eye disorders) | 1/6 | 0/26 | 0/28
Dysphagia (Gastrointestinal disorders) | 1/6 | 0/26 | 0/28
GLOSSODYNIA (Gastrointestinal disorders) | 1/6 | 0/26 | 0/28
SWOLLEN TONGUE (Gastrointestinal disorders) | 1/6 | 0/26 | 0/28
Pain (General disorders) | 0/6 | 1/26 | 2/28
CHEST DISCOMFORT (General disorders) | 0/6 | 2/26 | 2/28
PYREXIA (General disorders) | 2/6 | 4/26 | 2/28
ALLERGY TO ARTHROPOD BITE (Immune system disorders) | 0/6 | 2/26 | 0/28
NASAL VESTIBULITIS (Infections and infestations) | 1/6 | 0/26 | 0/28
RHINITIS (Infections and infestations) | 0/6 | 2/26 | 5/28
NASOPHARYNGITIS (Infections and infestations) | 1/6 | 2/26 | 4/28
FACE INJURY (Injury, poisoning and procedural complications) | 1/6 | 0/26 | 0/28
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1/6 | 0/26 | 0/28
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1/6 | 1/26 | 0/28
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1/6 | 3/26 | 1/28
DYSGEUSIA (Nervous system disorders) | 1/6 | 0/26 | 0/28
LETHARGY (Nervous system disorders) | 1/6 | 0/26 | 0/28
DIZZINESS (Nervous system disorders) | 1/6 | 1/26 | 0/28
HEADACHE (Nervous system disorders) | 4/6 | 15/26 | 12/28
SPUTUM DISCOLOURED (Respiratory, thoracic and mediastinal disorders) | 0/6 | 0/26 | 2/28
NASAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1/6 | 0/26 | 0/28
NASAL MUCOSAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 3/6 | 0/26 | 0/28
NASAL SEPTUM ULCERATION (Respiratory, thoracic and mediastinal disorders) | 2/6 | 0/26 | 0/28
UPPER AIRWAY OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 4/6 | 0/26 | 0/28
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 3/6 | 1/26 | 4/28
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1/6 | 1/26 | 4/28
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 1/6 | 1/26 | 0/28
COUGH (Respiratory, thoracic and mediastinal disorders) | 1/6 | 2/26 | 7/28
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 4/6 | 2/26 | 4/28
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 0/6 | 2/26 | 2/28
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 2/6 | 2/26 | 1/28
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4/6 | 3/26 | 2/28
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0/6 | 3/26 | 2/28
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0/6 | 4/26 | 4/28
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2/6 | 5/26 | 8/28
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2/6 | 0/26 | 1/28
RASH (Skin and subcutaneous tissue disorders) | 1/6 | 2/26 | 2/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between PI and Sponsor (AZ) or its agents that restricts the PI's right to discuss/publish trial results after the trial is completed. The PI agrees to collaborate in good faith with AZ with regards to content and formation of any publication or disclosure to be made by PI and to pay due consideration to opinions offered by AZ